CLINICAL TRIAL: NCT01089426
Title: Research Study of an Intravenous Fat Emulsion Comprised of Fish Oils (Omegaven) in the Treatment of Parenteral Nutrition (PN) Induced Liver Injury
Brief Title: Omegaven Treatment of Parenteral Nutrition (PN) Induced Liver Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Russell Merritt, Medical Director of Nutrition Support and Intestinal Rehabilitation, Children's Hospital Los Angeles
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCI-08-00127
Record Dates: First submitted 2010-03-15; First posted 2010-03-18 (Estimated); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Liver Injury
Keywords: Pediatric patients with Parenteral Nutrition (PN) induced Liver Injury
MeSH Terms: interventions — fish oil triglycerides; Administration, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Historical controls (Other): A subset of patients previously seen, who have had at least 2 consecutive direct bilirubin levels > 2 mg/dL, who depended on parenteral nutrition for at least 90 days after surgical therapy for congenital or acquired intestinal diseases
  Interventions: Other: Historical Controls
- Omegaven™ (Experimental)
  Interventions: Drug: Omegaven™

INTERVENTIONS:
Drug: Omegaven™ — 1 g/kg/d of Omegaven until discontinuation of PN
  Other Names: Highly refined fish oil for intravenous administration (10% Omegaven™)
  Arms: Omegaven™
Other: Historical Controls — Standard of Care
  Arms: Historical controls

SUMMARY:
This study examines the hypothesis that administering intravenous fish oil, in lieu of intravenous soybean oil, can ameliorate the progression of PN-associated cholestatic liver disease in pediatric patients with elevated direct bilirubin requiring PN for more than 30 days.

DETAILED DESCRIPTION:
In the United States, patients dependent upon parenteral nutrition (PN) receive parenteral fat emulsions composed of soybean oils. Lipids are necessary in PN dependent patients due to their high caloric value and essential fatty acid content. They have been implicated in predisposing patients to PN associated liver disease. Phytosterols such as those contained in soybean oils are thought to have a deleterious effect on biliary secretion.

Children requiring prolonged PN are at risk for developing PN associated liver disease. We hypothesize that although omega-6 fatty acid emulsions prevent fatty acid deficiency, they are not cleared in a manner similar to enteral chylomicrons and therefore accumulate in the liver and resulting in steatotic liver injury. We further hypothesize that a fat emulsion comprised of omega-3 fatty acids (i.e., fish oil) such as Omegaven™ would be beneficial in the management of steatotic liver injury by its inhibition of de novo lipogenesis, the reduction of arachidonic acid-derived inflammatory mediators, prevention of essential fatty acid deficiency through the presence of small amounts of arachidonic acid, and improved clearance of lipids from the serum. Animal studies have shown that IV fat emulsions (IFE) such as fish oil that are high in eicosapentaenic and docashexaaenoic acid reduce impairment of bile flow which is seen in cholestasis caused by conventional fat emulsions. Intravenous omega three fatty acids may be well tolerated and might reduce the inflammatory effect in the liver of prolonged PN exposure and could potentially reverse any hepatic dysfunction due to PN/IFE use. By administering Omegaven™ in place of conventional phytosterol/soybean fat emulsions we may reverse or prevent the progression of PN associated cholestasis and thus allow the patient to be maintained on adequate PN until they are able to ingest adequate nutrition enterally.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be parenteral nutrition dependent and are expected to require PN for at least another 30 days
* Patients must have parenteral nutrition associated liver disease (PNALD) as defined by having at least 2 consecutive direct bilirubins >2 mg/dl.

Exclusion Criteria:

* Pregnancy
* Other causes of liver disease
* Enrollment in any other clinical trial involving an investigational agent (unless approved by the designated physicians on the multidisciplinary team)
* Direct bilirubin < 2 mg/dl
* Allergy to any fish product, egg protein, and/or previous allergy to Omegaven
* Active coagulopathy characterized by on-going bleeding or acute need for clotting factor replacement such as FFP or cryoprecipitate to maintain homeostasis
* Impaired lipid metabolism as defined by serum Tg level >400 at time of initiation of Omegaven
* Unstable diabetes mellitus
* Recent stroke/embolism, not including catheter related thrombosis, which is a common complication of central venous catheter.
* Collapse and shock
* Undefined coma status
* Untreated infection at time of initiation of Omegaven
* Hemodynamic instability
* > 21 years of age

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2008-09; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Rate of reduction of direct bilirubin | normalization of direct bilirubin: an expected average of approximately 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Russell Merritt, M.D., PhD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Childrens Hospital Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Background] Dudrick SJ, Wilmore DW, Vars HM, Rhoads JE. Long-term total parenteral nutrition with growth, development, and positive nitrogen balance. Surgery. 1968 Jul;64(1):134-42. No abstract available. PMID 4968812
- [Background] Wilmore DW, Dudrick SJ. Growth and development of an infant receiving all nutrients exclusively by vein. JAMA. 1968 Mar 4;203(10):860-4. No abstract available. PMID 4965871
- [Background] Mullick FG, Moran CA, Ishak KG. Total parenteral nutrition: a histopathologic analysis of the liver changes in 20 children. Mod Pathol. 1994 Feb;7(2):190-4. PMID 8008742
- [Background] Freund HR. Abnormalities of liver function and hepatic damage associated with total parenteral nutrition. Nutrition. 1991 Jan-Feb;7(1):1-5; discussion 5-6. PMID 1802177
- [Background] Beath SV, Davies P, Papadopoulou A, Khan AR, Buick RG, Corkery JJ, Gornall P, Booth IW. Parenteral nutrition-related cholestasis in postsurgical neonates: multivariate analysis of risk factors. J Pediatr Surg. 1996 Apr;31(4):604-6. doi: 10.1016/s0022-3468(96)90507-2. PMID 8801324
- [Background] Greenberg GR, Wolman SL, Christofides ND, Bloom SR, Jeejeebhoy KN. Effect of total parenteral nutrition on gut hormone release in humans. Gastroenterology. 1981 May;80(5 pt 1):988-93. No abstract available. PMID 6781979
- [Background] Yeh SL, Chen WJ, Huang PC. Effects of L-glutamine on induced hepatosteatosis in rats receiving total parenteral nutrition. J Formos Med Assoc. 1995 Oct;94(10):593-9. PMID 8527958
- [Background] Kubota A, Yonekura T, Hoki M, Oyanagi H, Kawahara H, Yagi M, Imura K, Iiboshi Y, Wasa K, Kamata S, Okada A. Total parenteral nutrition-associated intrahepatic cholestasis in infants: 25 years' experience. J Pediatr Surg. 2000 Jul;35(7):1049-51. doi: 10.1053/jpsu.2000.7769. PMID 10917294
- [Background] Moss RL, Das JB, Ansari G, Raffensperger JG. Hepatobiliary dysfunction during total parenteral nutrition is caused by infusate, not the route of administration. J Pediatr Surg. 1993 Mar;28(3):391-6; discussion 396-7. doi: 10.1016/0022-3468(93)90238-g. PMID 8468653
- [Background] Helms RA, Christensen ML, Mauer EC, Storm MC. Comparison of a pediatric versus standard amino acid formulation in preterm neonates requiring parenteral nutrition. J Pediatr. 1987 Mar;110(3):466-70. doi: 10.1016/s0022-3476(87)80519-x. No abstract available. PMID 3102712
- [Background] Moss RL, Haynes AL, Pastuszyn A, Glew RH. Methionine infusion reproduces liver injury of parenteral nutrition cholestasis. Pediatr Res. 1999 May;45(5 Pt 1):664-8. doi: 10.1203/00006450-199905010-00009. PMID 10231861
- [Background] Meehan JJ, Georgeson KE. Prevention of liver failure in parenteral nutrition-dependent children with short bowel syndrome. J Pediatr Surg. 1997 Mar;32(3):473-5. doi: 10.1016/s0022-3468(97)90609-6. PMID 9094021
- [Background] Whalen GF, Shamberger RC, Perez-Atayde A, Folkman J. A proposed cause for the hepatic dysfunction associated with parenteral nutrition. J Pediatr Surg. 1990 Jun;25(6):622-6. doi: 10.1016/0022-3468(90)90348-d. PMID 2113578
- [Background] Zamir O, Nussbaum MS, Bhadra S, Subbiah MT, Rafferty JF, Fischer JE. Effect of enteral feeding on hepatic steatosis induced by total parenteral nutrition. JPEN J Parenter Enteral Nutr. 1994 Jan-Feb;18(1):20-5. doi: 10.1177/014860719401800120. PMID 8164298
- [Background] Kaminski DL, Adams A, Jellinek M. The effect of hyperalimentation on hepatic lipid content and lipogenic enzyme activity in rats and man. Surgery. 1980 Jul;88(1):93-100. No abstract available. PMID 6104363
- [Background] Hultin M, Carneheim C, Rosenqvist K, Olivecrona T. Intravenous lipid emulsions: removal mechanisms as compared to chylomicrons. J Lipid Res. 1995 Oct;36(10):2174-84. PMID 8576643
- [Background] Qi K, Al-Haideri M, Seo T, Carpentier YA, Deckelbaum RJ. Effects of particle size on blood clearance and tissue uptake of lipid emulsions with different triglyceride compositions. JPEN J Parenter Enteral Nutr. 2003 Jan-Feb;27(1):58-64. doi: 10.1177/014860710302700158. PMID 12549600
- [Background] Nestel PJ. Effects of N-3 fatty acids on lipid metabolism. Annu Rev Nutr. 1990;10:149-67. doi: 10.1146/annurev.nu.10.070190.001053. No abstract available. PMID 2200461
- [Background] Chen WJ, Yeh SL, Huang PC. Effects of fat emulsions with different fatty acid composition on plasma and hepatic lipids in rats receiving total parenteral nutrition. Clin Nutr. 1996 Feb;15(1):24-8. doi: 10.1016/s0261-5614(96)80257-3. PMID 16843991
- [Background] Yeh SL, Chen WJ, Huang PC. Effects of fish oil and safflower oil emulsions on diet-induced hepatic steatosis in rats receiving total parenteral nutrition. Clin Nutr. 1996 Apr;15(2):80-3. doi: 10.1016/s0261-5614(96)80024-0. PMID 16844003
- [Background] Kinsella JE, Lokesh B, Broughton S, Whelan J. Dietary polyunsaturated fatty acids and eicosanoids: potential effects on the modulation of inflammatory and immune cells: an overview. Nutrition. 1990 Jan-Feb;6(1):24-44; discussion 59-62. No abstract available. PMID 2135755
- [Background] Alwayn IP, Gura K, Nose V, Zausche B, Javid P, Garza J, Verbesey J, Voss S, Ollero M, Andersson C, Bistrian B, Folkman J, Puder M. Omega-3 fatty acid supplementation prevents hepatic steatosis in a murine model of nonalcoholic fatty liver disease. Pediatr Res. 2005 Mar;57(3):445-52. doi: 10.1203/01.PDR.0000153672.43030.75. Epub 2005 Jan 19. PMID 15659701
- [Background] Van Aerde JE, Duerksen DR, Gramlich L, Meddings JB, Chan G, Thomson AB, Clandinin MT. Intravenous fish oil emulsion attenuates total parenteral nutrition-induced cholestasis in newborn piglets. Pediatr Res. 1999 Feb;45(2):202-8. doi: 10.1203/00006450-199902000-00008. PMID 10022591
- [Background] Morlion BJ, Torwesten E, Lessire H, Sturm G, Peskar BM, Furst P, Puchstein C. The effect of parenteral fish oil on leukocyte membrane fatty acid composition and leukotriene-synthesizing capacity in patients with postoperative trauma. Metabolism. 1996 Oct;45(10):1208-13. doi: 10.1016/s0026-0495(96)90237-1. PMID 8843174
- [Background] Grimminger F, Fuhrer D, Papavassilis C, Schlotzer E, Mayer K, Heuer KU, Kiss L, Walmrath D, Piberhofer S, Lubbecke F, et al. Influence of intravenous n-3 lipid supplementation on fatty acid profiles and lipid mediator generation in a patient with severe ulcerative colitis. Eur J Clin Invest. 1993 Nov;23(11):706-15. doi: 10.1111/j.1365-2362.1993.tb01290.x. PMID 8307090
- [Background] Grimminger F, Mayser P, Papavassilis C, Thomas M, Schlotzer E, Heuer KU, Fuhrer D, Hinsch KD, Walmrath D, Schill WB, et al. A double-blind, randomized, placebo-controlled trial of n-3 fatty acid based lipid infusion in acute, extended guttate psoriasis. Rapid improvement of clinical manifestations and changes in neutrophil leukotriene profile. Clin Investig. 1993 Aug;71(8):634-43. doi: 10.1007/BF00184491. PMID 8219661
- [Background] Mayser P, Mrowietz U, Arenberger P, Bartak P, Buchvald J, Christophers E, Jablonska S, Salmhofer W, Schill WB, Kramer HJ, Schlotzer E, Mayer K, Seeger W, Grimminger F. Omega-3 fatty acid-based lipid infusion in patients with chronic plaque psoriasis: results of a double-blind, randomized, placebo-controlled, multicenter trial. J Am Acad Dermatol. 1998 Apr;38(4):539-47. doi: 10.1016/s0190-9622(98)70114-8. PMID 9555791
- [Background] Heller AR, Fischer S, Rossel T, Geiger S, Siegert G, Ragaller M, Zimmermann T, Koch T. Impact of n-3 fatty acid supplemented parenteral nutrition on haemostasis patterns after major abdominal surgery. Br J Nutr. 2002 Jan;87 Suppl 1:S95-101. doi: 10.1079/bjn2001462. PMID 11895160
- [Background] Gura KM, Parsons SK, Bechard LJ, Henderson T, Dorsey M, Phipatanakul W, Duggan C, Puder M, Lenders C. Use of a fish oil-based lipid emulsion to treat essential fatty acid deficiency in a soy allergic patient receiving parenteral nutrition. Clin Nutr. 2005 Oct;24(5):839-47. doi: 10.1016/j.clnu.2005.05.020. PMID 16029913
- [Background] Andorsky DJ, Lund DP, Lillehei CW, Jaksic T, Dicanzio J, Richardson DS, Collier SB, Lo C, Duggan C. Nutritional and other postoperative management of neonates with short bowel syndrome correlates with clinical outcomes. J Pediatr. 2001 Jul;139(1):27-33. doi: 10.1067/mpd.2001.114481. PMID 11445790